CLINICAL TRIAL: NCT07017712
Title: Sex Differences in Gastrointestinal Cancer Surgery
Acronym: SeDiGCS
Status: Completed | Type: Observational
Sponsor: Medizinische Hochschule Brandenburg Theodor Fontane (Other)
Responsible Party: Principal Investigator, Richard Hunger, Senior research assistant, Medizinische Hochschule Brandenburg Theodor Fontane
Other Study IDs: SeDiGCS
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-05

CONDITIONS: Sex; Gastrointestinal Cancers; Surgical Resection; Sex Differences
Keywords: Surgical Outcomes; Sex Differences; Surgical Otcomes Research
MeSH Terms: conditions — Coitus; Gastrointestinal Neoplasms | interventions — Proctectomy; Gastrectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Male patients
  Interventions: Procedure: Complex esophageal surgery for carcinoma; Procedure: Rectum resection for carcinoma; Procedure: Colon resection for carcinoma; Procedure: Pancreatic resection for carcinoma; Procedure: Gastric resection for carcinoma
- Female patients
  Interventions: Procedure: Complex esophageal surgery for carcinoma; Procedure: Rectum resection for carcinoma; Procedure: Colon resection for carcinoma; Procedure: Pancreatic resection for carcinoma; Procedure: Gastric resection for carcinoma

INTERVENTIONS:
Procedure: Complex esophageal surgery for carcinoma — Appropriate combination of ICD-10 code (C15, C16.0) and medical procedure code (5-423, 5-424, 5-425, 5-426, 5-427.0, 5-427.1, 5-438.0, 5-438.1, 5-438.x)
Procedure: Rectum resection for carcinoma — Appropriate combination of ICD-10 code (C19, C20, C218, D011, D012) and medical procedure code (5-484, 5-485)
Procedure: Colon resection for carcinoma — Appropriate combination of ICD-10 code (C18, D01.0) and medical procedure code (5-455, 5-456, 5-458)
Procedure: Pancreatic resection for carcinoma — Appropriate combination of ICD-10 code (C25, C24.1) and medical procedure code (5-524, 5-525.0, 5-525.1, 5-525.2, 5-525.x, 5-525.y, 5-528)
Procedure: Gastric resection for carcinoma — Appropriate combination of ICD-10 code (C16) and medical procedure code (5-436, 5-437, 5-438)

SUMMARY:
This study aims to investigate whether there are differences in surgical outcomes between male and female patients with gastrointestinal cancers (esophagus, colon, rectum, stomach, or pancreas). Previous research suggests that women may have worse outcomes after high-risk surgeries, such as heart or vascular procedures, but it is unclear if this applies to gastrointestinal cancer surgery. The study will analyze population based data from Germany to compare how often male and female patients died or died after the occurence of a surgical complication (failure to rescue) after surgery. The goal is to determine if biological sex influences surgical risks and recovery, which could help improve personalized care for cancer patients.

DETAILED DESCRIPTION:
DATA SOURCE

As database the German diagnosis-related group statistic (DRG statistic) will be queried. The dataset is provided by the German Federal Statistical Office. It includes standardized demographic information (age, sex), diagnostic codes (ICD-10-GM), procedural codes (OPS), and outcomes (mortality, length of stay, complications). Patients will be included if they underwent resection for one of the five specified cancers; exclusions applied for age <18 years, missing sex/age data, or non-matching diagnosis-procedure pairs.

OUTCOMES

Primary Endpoints:

Mortality: Death during the hospital stay. Failure-to-Rescue (FTR): Death among patients who developed postoperative complications (defined via appropriate ICD-10-GM/OPS codes)

Secondary Endpoints: 30-day mortality, complication rates, intensive care unit (ICU) admission, reoperation, and prolonged hospitalization (>75th percentile for procedure-specific stay). Failure to rescue rates of patients with extended medical treatment (eg. after reoperation, ICU admission, possibly in combination with a complication).

Adjustment Variables: Age, Elixhauser comorbidities (categorized using Quan's algorithm), admission type (elective/emergent), annual hospital procedure volume (to account for surgical expertise and routine), and year of surgery (to account for temporal trends).

Descriptive Analysis:

Data Validation: Checks will be performed to identify implausible values (e.g., age >120 years) or inconsistencies (e.g., mortality coded without complication for FTR analysis). Comorbidity Coding: Elixhauser comorbidities will be determined. Hospital Volume Metrics: Annual procedure volumes will be calculated to control for institutional expertise.

Statistical Analysis Plan As primary analysis, multivariable logistic regression models will be calculated that assessed sex differences in mortality/FTR, adjusting for covariates (age, individual Elixhauser comorbidities, hospital volume, and admission type, year of surgery). Adjusted odds ratios (aORs) and adjusted risk differences (aRD) with 95% confidence intervals (CIs) will be reported.

Subgroup / Sensitivity Analyses:

To ensure robustness of results multiple sensitivity analyses will be performed. These include subgroup analysis where tha analysis will be perfomed by startified groups:

1. by admission type (elective vs. emergent),
2. by comorbidity burden (≤3 vs. >4 Elixhauser conditions), and
3. by hospital volume (above/below median).

REPORTING

Descriptive/Univariable analysis:

This study will report descriptively baseline patient characteristics and compare the charachteristics between male and female patients. Tests will be selected according to variable type (categorical vs. continuous) and type of distribution (normal vs non-normal distributed).

Observed outcome rates will be reported and compared between male and female patients. Observed risk differences and risk ratios will be calculated.

Multivariable analysis:

Results of the multivariable logistic regressions will be reported as adjusted risk differences and/or adjusted risk ratios. Appropriate figures will be produced to communicate the results. Sensitivity analyses stratified by admission type, comorbidity burden, and hospital volume will reinforce the robustness of these results.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old at the time of the operation
* Rectum resection for carcinoma (ICD-10: C19, C20, C218, D01.1, D01.2) and appropriate resection procedure (5-484, 5-485)
* Colon resection for carcinoma (ICD-10: C18, D01.0) and appropriate resection procedure (5-455, 5-456, 5-458)
* Complex esophageal surgery for carcinoma (ICD-10: C15, C16.0) and appropriate resection procedure (5-423, 5-424, 5-425, 5-426, 5-427.0, 5-427.1, 5-438.0, 5-438.1, 5-438.x)
* Pancreatic resection for carcinoma (ICD-10: C25, C24.1) and appropriate resection procedure (5-524, 5-525.0, 5-525.1, 5-525.2, 5-525.x, 5-525.y, 5-528)
* Gastric resection for carcinoma (ICD-10: C16) and appropriate resection procedure (5-436, 5-437, 5-438)

Exclusion Criteria:

* missing data for age and/or sex
* implausible combination of diagnosis and resection procedure (eg. a patient with a gastrectomy but without appropriate ICD-10 diagnosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population based study. Principally all patients that underwent any of the described procedures in an German hospital are included in the dataset.
Sampling Method: Non-Probability Sample
Enrollment: 870754 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Mortality rate | Up to 90 days postoperatively
  Proportion of patients that died after surgical intervention
Failure to rescue | Up to 90 days postoperatively
  Proportion of patients that died after the occurence of a postoperative complication

SECONDARY OUTCOMES:
Complication rate | Up to 90 days postoperatively
  Folloing individual comorbidities are considered:
  Acute myocardial infarction Acute pulmonary embolism Pulmonary insufficiency Sepsis Shock during or resulting from a procedure Shock due to anaesthesia Toxic shock Septic shock Anaphylactic shock Renal failure Haemorrhage Accidental puncture and laceration during a procedure Disruption of operation wound Infection Foreign body accidentally left in body cavity or operation wound following a procedure Acute reaction to foreign substance accidentally left during a procedure Vascular complications following a procedure Other complications of procedures Pancreatoduodenal fistula Peritonitis Anastomotic insufficiency Postoperative bowel occlusion Blood transfusion Other specified complications of surgical and medical care Complication of surgical and medical care, unspecified
Reoperation rate | Up to 90 days postoperatively
  Reoperation during the same hospital stay of the index operation. Identified using the following medical procedure code: 5-983.
Intensive Care Unit admission | Up to 90 days postoperatively
  Postoperative admission to the Intensive Care Unit
Prolonged Lenght of Stay | Up to 90 days postoperatively
  Length of stay above the 75. percentile of all patients with the same diagnosis / procedure combination
Failure to rescue | Up to 90 days postoperatively
  Proportion of patients that died after the occurence of any of the other secondary outcome measures

IPD SHARING:
Plan to Share IPD: No
The dissemination of Diagnosis-Related Group (DRG) statistics is not a viable option due to the centralised management of such data by the Federal Statistical Office of Germany, which restricts accessibility and analysis to remote mechanisms.